CLINICAL TRIAL: NCT05050812
Title: The Grounded Brain: How Sleeping Grounded (Earthing) Affects Cognition and Personal Perceptions in Participants With Mild Cognitive Impairment Due to Alzheimer's Disease (MCI/AD)
Brief Title: The Grounded Brain: How Sleeping Grounded Affects Memory and Perceptions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: California Institute of Integral Studies (Other)
Responsible Party: Principal Investigator, Patrice F. Jones, Student Researcher, California Institute of Integral Studies
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PFJ001
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Mild Cognitive Impairment; Chronic Inflammation
Keywords: Earthing; systemic chronic inflammation; grounding; SCI; immune system; sleep quality; mood; pain; well-being; mild cognitive impairment due to Alzheimer's disease; MCI; glucocorticoid resistance; neurodegenerative; Cogstate Cognitive Brief Battery; Cogstate CBB
MeSH Terms: conditions — Cognitive Dysfunction; Sleep Initiation and Maintenance Disorders; Pain; Glucocorticoid Receptor Deficiency

STUDY DESIGN:
Intervention Model Description: An interventional, single-group method that lacks random assignment and has no control group but does provide baseline and post-intervention testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Grounded (Experimental): All participants will sleep on a grounding mat for at least six hours per 24-hour period.
  Interventions: Device: grounding mat

INTERVENTIONS:
Device: grounding mat — Participants will sleep on an Earthing Elite sleep mat produced and sold by Earthing.com
  Other Names: Earthing mat

SUMMARY:
Grounding (Earthing) refers to the practice of contacting the Earth or a properly installed grounding mat with the body. Previous studies on grounding have shown positive effects body-wide inflammation, acute and chronic pain, and immune system response. Prior studies on the inflammatory process of mild cognitive impairment due to Alzheimer's disease, Alzheimer's disease, and some other dementias have shown connections between immune system dysregulation, inflammatory markers, and severe disease progression. Finding ways to mitigate or turn off the inflammatory response is key to treating mild cognitive impairment due to Alzheimer's disease. The purpose of this study is to evaluate the effects of sleeping grounded on cognition and personal perceptions in participants with a diagnosis of mild cognitive impairment due to Alzheimer's disease as evidenced by a battery of assessments using Cogstate's Cognitive Brief Battery and a qualitative questionnaire. We hypothesize that assessment scores will improve with grounding and that perceptions will positively correlate with an increase in scores. Modulation of risk factors like glucocorticoid resistance, SCI, and immune system dysfunction through grounding may lead to an accessible, natural technique for neurodegenerative disease prevention or treatment.

DETAILED DESCRIPTION:
Grounding (Earthing) refers to the practice of contacting the Earth or a properly installed grounding mat with the body. Previous studies on grounding have shown positive effects on diurnal cortisol regulation, systemic chronic inflammation (SCI), immune system response, acute and chronic pain, mood, vagal tone, blood viscosity, blood flow, recovery from muscle strain and damage, and prevention or mitigation of chronic inflammatory and autoimmune diseases. Prior studies on the inflammatory process of mild cognitive impairment due to Alzheimer's disease, Alzheimer's disease, and some other dementias have shown connections between immune system dysregulation, inflammatory markers, and severe disease progression. The purpose of this study is to evaluate the effects of sleeping grounded on cognition and personal perceptions in participants with a diagnosis of mild cognitive impairment due to Alzheimer's disease (MCI/AD) as evidenced by a battery of tests using the Cogstate platform's Cognitive Brief Battery (CBB) and a qualitative questionnaire to detect any correlations to the participant's perceptions of sleep quality, mood, pain, and overall well-being.

This study will both fulfill the requirement for a Bachelor of Science in Psychology and lay the foundation for further research into grounding and neurodegenerative diseases. My senior research project methodology is a mixed methods research design with a triangulation convergence, since I'll be concurrently collecting, analyzing, and evaluating the results of the quantitative and qualitative measurements before comparing, integrating, and interpreting the outcomes.

I have three hypotheses. First, I hypothesize that sleeping while grounded will result in improved scores on the Cogstate battery of tests given at baseline and weekly for three weeks. Second, I hypothesize that sleeping while grounded will result in positive perceptions regarding sleep quality, mood, pain, and overall well-being. Finally, I hypothesize that improved Cogstate scores will positively correlate with perceptions of sleep quality, mood, and overall well-being and negatively correlate with pain. The independent variable is the intervention (grounded sleeping mat), and the dependent variables are the three measurements of cognition (memory, working memory, and processing speed) and the qualitative questionnaire to evaluate how the participants feel about their sleep quality, mood, pain, and overall well-being.

The target population for this study will be adults aged 55 and up (N=8) with a current diagnosis of MCI/AD who meet the inclusion and exclusion criteria. I will employ a mixed methods research design that includes statistical analysis of empirical data and a qualitative questionnaire. I will use a triangulation convergence, since I'll be concurrently collecting, analyzing, and evaluating the results of the quantitative and qualitative measurements before comparing, integrating, and interpreting the outcomes. First, I will look at the percentage of change in each testing area from week to week and calculate the statistical significance (p < .01) of any changes. Second, I will calculate the mean of all the test scores per day (baseline and weekly X 3) to obtain a general cognition score which I will also use to calculate statistical significance (p < .01) of changes over time. Third, I will perform a simple linear regression analysis to determine if a correlation exists between the intervention and the cognition scores after baseline. Finally, I will perform an analysis of the qualitative questionnaire using in vivo coding to determine if any correlations exist between the cognition scores and personal perceptions. For this study, I will interpret the results based on changes in test scores over time, changes in general cognition scores over time, and positive/negative correlations of the personal perceptions and cognition scores.

Each participant will receive an Earthing Elite™ sleep mat kit which they get to keep. The sleeping mat will be installed wherever the participant sleeps (bed or recliner), and I will ensure that the mat is properly attached to the grounding plug and confirm grounding using a multimeter with two terminal leads, a cord with alligator clips on both ends, an Earthing coil cord, and an outlet checker. This procedure will show body voltage prior to grounding and while grounding to confirm that the setup is working and that body voltage has been neutralized. I will return for repeat assessments after one week, two weeks, and three weeks at which time I will verify that the system is still working properly.

All computerized testing will consist of the following assessments on the Cogstate platform: 1) Detection test (psychomotor function); 2) Identification test (attention); 3) One Card Learning test (visual learning); and 4) One Back test (working memory). The personal perceptions qualitative questionnaire will consist of several open-ended and scaled questions designed to assess how the participants perceive various subjective areas such as sleep quality, pain, mood, and overall well-being. Each participant will complete the questionnaire first before completing the computerized cognition assessments.

Modulation of risk factors like glucocorticoid resistance, SCI, and immune system dysfunction through grounding may lead to an accessible, natural technique for neurodegenerative disease prevention or treatment.

ELIGIBILITY:
Inclusion Criteria:

* All approved participants must

  1. Be at least 55 years of age; all genders and ethnicities;
  2. Have English as their primary language or be able to speak, read, and write English fluently; As this is a vulnerable population, this investigator must be able to evaluate understanding and cannot reliably do that with someone who is not fluent in English;
  3. Have a current diagnosis of mild cognitive impairment due to Alzheimer's disease made by a medical doctor;
  4. Be able to spend at least 6 hours per 24-hour period sleeping or resting on the grounded mat;
  5. Be able to legally consent to participating in this study;
  6. Agree to allow the researcher to come into their home to setup the equipment and administer the tests;
  7. Be able to see well enough to use a laptop to complete electronic testing;
  8. Be alert and oriented X 4 based on initial verbal screening and in-person visits;
  9. Reside in or around the Greater Austin, Texas, area/Central Texas area;
  10. Sleep in a dwelling that is grounded.

Exclusion Criteria:

* All approved participants must

  1. Not have a diagnosis or conversion to AD or any other type of memory disorder before or during the study period including but not limited to dementia, Lewy body disease, Creutzfeldt-Jakob disease, Parkinson's disease, Huntington's disease, vascular cognitive impairment, frontotemporal dementias, primary progressive aphasia, autoimmune encephalopathy, and normal pressure hydrocephalus;
  2. Not have a diagnosis of stable MCI;
  3. Not have any prior diagnosis of traumatic brain injury;
  4. Not have any history of grounding consistently for more than 60 minutes/day in the past year. This includes natural methods and the use of any grounding devices;
  5. Not have any in-the-moment assessment that leads the investigator to believe that the participant is not fully aware or does not understand what is being asked of them. Again, this is a vulnerable population, and I will exclude or cut any participant who shows signs of confusion;
  6. Not be taking or have taken in the previous 30 days any of the following medications:

     1. daily anti-inflammatories, prescription or over the counter;
     2. blood pressure medications (anti-hypertensives);
     3. blood thinners (anti-coagulants);

     e. glucose control medications; f. thyroid medications; g. anti-convulsive medications (no matter the diagnosis); h. any type of monoclonal antibody; i. any type of immunosuppressive, including steroids; j. any type of immunomodulator.
  7. Inability to answer the questions in the initial screening interview;
  8. Inability to follow instructions.

A Note About Medications and Grounding:

Earthing has been proven to reduce inflammation, thin the blood, lower blood pressure, lower and better regulate glucose levels, and improve thyroid function. While all those things are generally sought after, there could be dire consequences if a participant is on a medication to correct any of those conditions, so in the interest of safety, exclusion based on certain medications is necessary. In that same vein, if any participant must begin a medication during the study period, that participant will be disqualified in the interest of safety.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Baseline Psychomotor Function Score | Baseline
  In this simple reaction time Detection test, a playing card is presented face-down in the center of the screen. After a random interval, the card will turn over so that is it face-up (revealing a Joker card - this same card is used throughout the test). The subject is asked to press the "YES" button as soon as the card turns face-up. Assessed at baseline then weekly for three weeks.
Week 1 Psychomotor Function Score | Week 1
  In this simple reaction time Detection test, a playing card is presented face-down in the center of the screen. After a random interval, the card will turn over so that is it face-up (revealing a Joker card - this same card is used throughout the test). The subject is asked to press the "YES" button as soon as the card turns face-up. Assessed at baseline then weekly for three weeks.
Week 2 Psychomotor Function Score | Week 2
  In this simple reaction time Detection test, a playing card is presented face-down in the center of the screen. After a random interval, the card will turn over so that is it face-up (revealing a Joker card - this same card is used throughout the test). The subject is asked to press the "YES" button as soon as the card turns face-up. Assessed at baseline then weekly for three weeks.
Week 3 Psychomotor Function Score | Week 3
  In this simple reaction time Detection test, a playing card is presented face-down in the center of the screen. After a random interval, the card will turn over so that is it face-up (revealing a Joker card - this same card is used throughout the test). The subject is asked to press the "YES" button as soon as the card turns face-up. Assessed at baseline then weekly for three weeks.
Change from Baseline to Week 3 Psychomotor Function Score | Change from baseline to week 3
  In this simple reaction time Detection test, a playing card is presented face-down in the center of the screen. After a random interval, the card will turn over so that is it face-up (revealing a Joker card - this same card is used throughout the test). The subject is asked to press the "YES" button as soon as the card turns face-up. Assessed at baseline then weekly for three weeks. Change = (Week 3 Psychomotor Function Score - Baseline Psychomotor Function Score).
Baseline Attention Score | Baseline
  In this choice reaction time Identification test, a playing card is presented face-down in the center of the screen. After a random interval, the card will turn over so that is it face-up. Either a red Joker card or black Joker card will be revealed. As soon as the card turns face-up, the subject decides whether the card displayed is red. If the card is red, the subject should press the "YES" button, if it is not red, they should press "NO". Assessed at baseline then weekly for three weeks.
Week 1 Attention Score | Week 1
  In this choice reaction time Identification test, a playing card is presented face-down in the center of the screen. After a random interval, the card will turn over so that is it face-up. Either a red Joker card or black Joker card will be revealed. As soon as the card turns face-up, the subject decides whether the card displayed is red. If the card is red, the subject should press the "YES" button, if it is not red, they should press "NO". Assessed at baseline then weekly for three weeks.
Week 2 Attention Score | Week 2
  In this choice reaction time Identification test, a playing card is presented face-down in the center of the screen. After a random interval, the card will turn over so that is it face-up. Either a red Joker card or black Joker card will be revealed. As soon as the card turns face-up, the subject decides whether the card displayed is red. If the card is red, the subject should press the "YES" button, if it is not red, they should press "NO". Assessed at baseline then weekly for three weeks.
Week 3 Attention Score | Week 3
  In this choice reaction time Identification test, a playing card is presented face-down in the center of the screen. After a random interval, the card will turn over so that is it face-up. Either a red Joker card or black Joker card will be revealed. As soon as the card turns face-up, the subject decides whether the card displayed is red. If the card is red, the subject should press the "YES" button, if it is not red, they should press "NO". Assessed at baseline then weekly for three weeks.
Change from Baseline to Week 3 Attention Score | Baseline to week 4
  In this choice reaction time Identification test, a playing card is presented face-down in the center of the screen. After a random interval, the card will turn over so that is it face-up. Either a red Joker card or black Joker card will be revealed. As soon as the card turns face-up, the subject decides whether the card displayed is red. If the card is red, the subject should press the "YES" button, if it is not red, they should press "NO". Assessed at baseline then weekly for three weeks. Change = (Week 3 Attention Score - Baseline Attention Score).
Baseline Visual Learning Score | Baseline
  In this pattern separation One Card Learning test, a playing card is presented face-down in the center of the screen. After a random interval, the card will turn over so that is it face-up. A regular playing card from a French deck is revealed. As soon as the card turns face-up, the subject must decide whether the current card has been seen before in the test. The subject should press the "YES" button if they have seen the card before in the test, or "NO" if they have not. Assessed at baseline then weekly for three weeks.
Week 1 Visual Learning Score | Week 1
  In this pattern separation One Card Learning test, a playing card is presented face-down in the center of the screen. After a random interval, the card will turn over so that is it face-up. A regular playing card from a French deck is revealed. As soon as the card turns face-up, the subject must decide whether the current card has been seen before in the test. The subject should press the "YES" button if they have seen the card before in the test, or "NO" if they have not. Assessed at baseline then weekly for three weeks.
Week 2 Visual Learning Score | Week 2
  In this pattern separation One Card Learning test, a playing card is presented face-down in the center of the screen. After a random interval, the card will turn over so that is it face-up. A regular playing card from a French deck is revealed. As soon as the card turns face-up, the subject must decide whether the current card has been seen before in the test. The subject should press the "YES" button if they have seen the card before in the test, or "NO" if they have not. Assessed at baseline then weekly for three weeks.
Week 3 Visual Learning Score | Week 3
  In this pattern separation One Card Learning test, a playing card is presented face-down in the center of the screen. After a random interval, the card will turn over so that is it face-up. A regular playing card from a French deck is revealed. As soon as the card turns face-up, the subject must decide whether the current card has been seen before in the test. The subject should press the "YES" button if they have seen the card before in the test, or "NO" if they have not. Assessed at baseline then weekly for three weeks.
Change from Baseline to Week 3 Visual Learning Score | Baseline to Week 3
  In this pattern separation One Card Learning test, a playing card is presented face-down in the center of the screen. After a random interval, the card will turn over so that is it face-up. A regular playing card from a French deck is revealed. As soon as the card turns face-up, the subject must decide whether the current card has been seen before in the test. The subject should press the "YES" button if they have seen the card before in the test, or "NO" if they have not. Assessed at baseline then weekly for three weeks. Change = (Week 3 Visual Learning Score - Baseline Visual Learning Score).
Baseline Working Memory Score | Baseline
  In this N-back One Back test, a playing card is presented face-down in the center of the screen. After a random interval, the card will turn over so that is it face-up. A regular playing card from a French deck is revealed. As soon as the card turns face-up, the subject must decide whether the current card is the same as the previous card. The subject should press the "YES" button if the current card is the same as the one presented immediately before it, or "NO" if it is not the same. Assessed at baseline and weekly for three weeks.
Week 1 Working Memory Score | Week 1
  In this N-back One Back test, a playing card is presented face-down in the center of the screen. After a random interval, the card will turn over so that is it face-up. A regular playing card from a French deck is revealed. As soon as the card turns face-up, the subject must decide whether the current card is the same as the previous card. The subject should press the "YES" button if the current card is the same as the one presented immediately before it, or "NO" if it is not the same. Assessed at baseline and weekly for three weeks.
Week 2 Working Memory Score | Week 2
  In this N-back One Back test, a playing card is presented face-down in the center of the screen. After a random interval, the card will turn over so that is it face-up. A regular playing card from a French deck is revealed. As soon as the card turns face-up, the subject must decide whether the current card is the same as the previous card. The subject should press the "YES" button if the current card is the same as the one presented immediately before it, or "NO" if it is not the same. Assessed at baseline and weekly for three weeks.
Week 3 Working Memory Score | Week 3
  In this N-back One Back test, a playing card is presented face-down in the center of the screen. After a random interval, the card will turn over so that is it face-up. A regular playing card from a French deck is revealed. As soon as the card turns face-up, the subject must decide whether the current card is the same as the previous card. The subject should press the "YES" button if the current card is the same as the one presented immediately before it, or "NO" if it is not the same. Assessed at baseline and weekly for three weeks.
Change from Baseline to Week 3 Working Memory Score | Baseline and Week 3
  In this N-back One Back test, a playing card is presented face-down in the center of the screen. After a random interval, the card will turn over so that is it face-up. A regular playing card from a French deck is revealed. As soon as the card turns face-up, the subject must decide whether the current card is the same as the previous card. The subject should press the "YES" button if the current card is the same as the one presented immediately before it, or "NO" if it is not the same. Assessed at baseline and weekly for three weeks. Change = (Week 3 Working Memory Score - Baseline Working Memory Score).
Baseline Sleep Quality Score | Baseline
  The Personal Perceptions Questionnaire is a self-designed instrument assessing a participant's perception about their average sleep quality, mood, pain, and well-being over the past 7 days. One question is open-ended and uses in vivo coding to create a score about sleep quality while the second question about sleep quality is scaled. Possible scores range from 0 (worst sleep quality) to 10 (best sleep quality).
Week 1 Sleep Quality Score | Week 1
  The Personal Perceptions Questionnaire is a self-designed instrument assessing a participant's perception about their average sleep quality, mood, pain, and well-being over the past 7 days. One question is open-ended and uses in vivo coding to create a score about sleep quality while the second question about sleep quality is scaled. Possible scores range from 0 (worst sleep quality) to 10 (best sleep quality).
Week 2 Sleep Quality Score | Week 2
  The Personal Perceptions Questionnaire is a self-designed instrument assessing a participant's perception about their average sleep quality, mood, pain, and well-being over the past 7 days. One question is open-ended and uses in vivo coding to create a score about sleep quality while the second question about sleep quality is scaled. Possible scores range from 0 (worst sleep quality) to 10 (best sleep quality).
Week 3 Sleep Quality Score | Week 3
  The Personal Perceptions Questionnaire is a self-designed instrument assessing a participant's perception about their average sleep quality, mood, pain, and well-being over the past 7 days. One question is open-ended and uses in vivo coding to create a score about sleep quality while the second question about sleep quality is scaled. Possible scores range from 0 (worst sleep quality) to 10 (best sleep quality).
Change from Baseline to Week 3 Sleep Quality Score | Week 3
  The Personal Perceptions Questionnaire is a self-designed instrument assessing a participant's perception about their average sleep quality, mood, pain, and well-being over the past 7 days. One question is open-ended and uses in vivo coding to create a score about sleep quality while the second question about sleep quality is scaled. Possible scores range from 0 (worst sleep quality) to 10 (best sleep quality). Change = (Week 3 Sleep Quality Score - Baseline Sleep Quality Score).
Baseline Pain Score | Baseline
  The Personal Perceptions Questionnaire is a self-designed instrument assessing a participant's perception about their average sleep quality, mood, pain, and well-being over the past 7 days. One question is open-ended and uses in vivo coding to create a score about pain while the second question about pain is scaled. Possible scores range from 0 (no pain) to 10 (worst pain).
Week 1 Pain Score | Week 1
  The Personal Perceptions Questionnaire is a self-designed instrument assessing a participant's perception about their average sleep quality, mood, pain, and well-being over the past 7 days. One question is open-ended and uses in vivo coding to create a score about pain while the second question about pain is scaled. Possible scores range from 0 (no pain) to 10 (worst pain).
Week 2 Pain Score | Week 2
  The Personal Perceptions Questionnaire is a self-designed instrument assessing a participant's perception about their average sleep quality, mood, pain, and well-being over the past 7 days. One question is open-ended and uses in vivo coding to create a score about pain while the second question about pain is scaled. Possible scores range from 0 (no pain) to 10 (worst pain).
Week 3 Pain Score | Week 3
  The Personal Perceptions Questionnaire is a self-designed instrument assessing a participant's perception about their average sleep quality, mood, pain, and well-being over the past 7 days. One question is open-ended and uses in vivo coding to create a score about pain while the second question about pain is scaled. Possible scores range from 0 (no pain) to 10 (worst pain).
Change from Baseline to Week 3 Pain Score | Baseline to Week 3
  The Personal Perceptions Questionnaire is a self-designed instrument assessing a participant's perception about their average sleep quality, mood, pain, and well-being over the past 7 days. One question is open-ended and uses in vivo coding to create a score about pain while the second question about pain is scaled. Possible scores range from 0 (no pain) to 10 (worst pain).
Baseline Mood Score | Baseline
  The Personal Perceptions Questionnaire is a self-designed instrument assessing a participant's perception about their average sleep quality, mood, pain, and well-being over the past 7 days. One question is open-ended and uses in vivo coding to create a score about mood while the second question about mood is scaled. Possible scores range from 0 (worst mood) to 10 (best mood).
Week 1 Mood Score | Week 1
  The Personal Perceptions Questionnaire is a self-designed instrument assessing a participant's perception about their average sleep quality, mood, pain, and well-being over the past 7 days. One question is open-ended and uses in vivo coding to create a score about mood while the second question about mood is scaled. Possible scores range from 0 (worst mood) to 10 (best mood).
Week 2 Mood Score | Week 2
  The Personal Perceptions Questionnaire is a self-designed instrument assessing a participant's perception about their average sleep quality, mood, pain, and well-being over the past 7 days. One question is open-ended and uses in vivo coding to create a score about mood while the second question about mood is scaled. Possible scores range from 0 (worst mood) to 10 (best mood).
Week 3 Mood Score | Week 3
  The Personal Perceptions Questionnaire is a self-designed instrument assessing a participant's perception about their average sleep quality, mood, pain, and well-being over the past 7 days. One question is open-ended and uses in vivo coding to create a score about mood while the second question about mood is scaled. Possible scores range from 0 (worst mood) to 10 (best mood).
Change from Baseline to Week 3 Mood Score | Baseline to Week 3
  The Personal Perceptions Questionnaire is a self-designed instrument assessing a participant's perception about their average sleep quality, mood, pain, and well-being over the past 7 days. One question is open-ended and uses in vivo coding to create a score about mood while the second question about mood is scaled. Possible scores range from 0 (worst mood) to 10 (best mood).
Baseline Overall Well-Being Score | Baseline
  The Personal Perceptions Questionnaire is a self-designed instrument assessing a participant's perception about their average sleep quality, mood, pain, and well-being over the past 7 days. One question is open-ended and uses in vivo coding to create a score about overall well-being while the second question about overall well-being is scaled. Possible scores range from 0 (worst overall well-being) to 10 (best overall well-being).
Week 1 Overall Well-Being Score | Week 1
  The Personal Perceptions Questionnaire is a self-designed instrument assessing a participant's perception about their average sleep quality, mood, pain, and well-being over the past 7 days. One question is open-ended and uses in vivo coding to create a score about overall well-being while the second question about overall well-being is scaled. Possible scores range from 0 (worst overall well-being) to 10 (best overall well-being).
Week 2 Overall Well-Being Score | Week 2
  The Personal Perceptions Questionnaire is a self-designed instrument assessing a participant's perception about their average sleep quality, mood, pain, and well-being over the past 7 days. One question is open-ended and uses in vivo coding to create a score about overall well-being while the second question about overall well-being is scaled. Possible scores range from 0 (worst overall well-being) to 10 (best overall well-being).
Week 3 Overall Well-Being Score | Week 3
  The Personal Perceptions Questionnaire is a self-designed instrument assessing a participant's perception about their average sleep quality, mood, pain, and well-being over the past 7 days. One question is open-ended and uses in vivo coding to create a score about overall well-being while the second question about overall well-being is scaled. Possible scores range from 0 (worst overall well-being) to 10 (best overall well-being).
Change from Baseline to Week 3 Overall Well-Being Score | Baseline to Week 3
  The Personal Perceptions Questionnaire is a self-designed instrument assessing a participant's perception about their average sleep quality, mood, pain, and well-being over the past 7 days. One question is open-ended and uses in vivo coding to create a score about overall well-being while the second question about overall well-being is scaled. Possible scores range from 0 (worst overall well-being) to 10 (best overall well-being).

SECONDARY OUTCOMES:
Correlation of Change in Psychomotor Function Score and Sleep Quality Score from Baseline to Week 3 | Baseline to Week 3
  Using simple regression to assess Baseline to Week 3 change in Psychomotor Function Score and whether that change positively or negatively correlates to the Change from Baseline to Week 3 Sleep Quality Score.
Correlation of Change in Psychomotor Function Score and Pain Score from Baseline to Week 3 | Baseline to Week 3
  Using simple regression to assess Baseline to Week 3 change in Psychomotor Function Score and whether that change positively or negatively correlates to the Change from Baseline to Week 3 Pain Score.
Correlation of Change in Psychomotor Function Score and Mood Score from Baseline to Week 3 | Baseline to Week 3
  Using simple regression to assess Baseline to Week 3 change in Psychomotor Function Score and whether that change positively or negatively correlates to the Change from Baseline to Week 3 Mood Score.
Correlation of Change in Psychomotor Function Score and Overall Well-Being Score from Baseline to Week 3 | Baseline to Week 3
  Using simple regression to assess Baseline to Week 3 change in Psychomotor Function Score and whether that change positively or negatively correlates to the Change from Baseline to Week 3 Overall Well-Being Score.
Correlation of Change in Attention Score and Sleep Quality Score from Baseline to Week 3 | Baseline to Week 3
  Using simple regression to assess Baseline to Week 3 change in Attention Score and whether that change positively or negatively correlates to the Change from Baseline to Week 3 Sleep Quality Score.
Correlation of Change in Attention Score and Pain Score from Baseline to Week 3 | Baseline to Week 3
  Using simple regression to assess Baseline to Week 3 change in Attention Score and whether that change positively or negatively correlates to the Change from Baseline to Week 3 Pain Score.
Correlation of Change in Attention Score and Mood Score from Baseline to Week 3 | Baseline to Week 3
  Using simple regression to assess Baseline to Week 3 change in Attention Score and whether that change positively or negatively correlates to the Change from Baseline to Week 3 Mood Score.
Correlation of Change in Attention Score and Overall Well-Being Score from Baseline to Week 3 | Baseline to Week 3
  Using simple regression to assess Baseline to Week 3 change in Attention Score and whether that change positively or negatively correlates to the Change from Baseline to Week 3 Overall Well-Being Score.
Correlation of Change in Visual Learning Score and Sleep Quality Score from Baseline to Week 3 | Baseline to Week 3
  Using simple regression to assess Baseline to Week 3 change in Visual Learning Score and whether that change positively or negatively correlates to the Change from Baseline to Week 3 Sleep Quality Score.
Correlation of Change in Visual Learning Score and Pain Score from Baseline to Week 3 | Baseline to Week 3
  Using simple regression to assess Baseline to Week 3 change in Visual Learning Score and whether that change positively or negatively correlates to the Change from Baseline to Week 3 Pain Score.
Correlation of Change in Visual Learning Score and Mood Score from Baseline to Week 3 | Baseline to Week 3
  Using simple regression to assess Baseline to Week 3 change in Visual Learning Score and whether that change positively or negatively correlates to the Change from Baseline to Week 3 Mood Score.
Correlation of Change in Visual Learning Score and Overall Well-Being Score from Baseline to Week 3 | Baseline to Week 3
  Using simple regression to assess Baseline to Week 3 change in Visual Learning Score and whether that change positively or negatively correlates to the Change from Baseline to Week 3 Overall Well-Being Score.
Correlation of Change in Working Memory Score and Sleep Quality Score from Baseline to Week 3 | Baseline to Week 3
  Using simple regression to assess Baseline to Week 3 change in Working Memory Score and whether that change positively or negatively correlates to the Change from Baseline to Week 3 Sleep Quality Score.
Correlation of Change in Working Memory Score and Pain Score from Baseline to Week 3 | Baseline to Week 3
  Using simple regression to assess Baseline to Week 3 change in Working Memory Score and whether that change positively or negatively correlates to the Change from Baseline to Week 3 Pain Score.
Correlation of Change in Working Memory Score and Mood Score from Baseline to Week 3 | Baseline to Week 3
  Using simple regression to assess Baseline to Week 3 change in Working Memory Score and whether that change positively or negatively correlates to the Change from Baseline to Week 3 Mood Score.
Correlation of Change in Working Memory Score and Overall Well-Being Score from Baseline to Week 3 | Baseline to Week 3
  Using simple regression to assess Baseline to Week 3 change in Working Memory Score and whether that change positively or negatively correlates to the Change from Baseline to Week 3 Overall Well-Being Score.

CONTACTS AND LOCATIONS:
Overall Officials: Patrice F Jones, CPC, Principal Investigator — California Institute of Integral Studies; Anne Huffman, PhD, Study Director — California Institute of Integral Studies

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bostrom G, Freyhult E, Virhammar J, Alcolea D, Tumani H, Otto M, Brundin RM, Kilander L, Lowenmark M, Giedraitis V, Lleo A, von Arnim CAF, Kultima K, Ingelsson M. Different Inflammatory Signatures in Alzheimer's Disease and Frontotemporal Dementia Cerebrospinal Fluid. J Alzheimers Dis. 2021;81(2):629-640. doi: 10.3233/JAD-201565. PMID 33814444
- [Result] Brown D, Chevalier G, Hill M. Pilot study on the effect of grounding on delayed-onset muscle soreness. J Altern Complement Med. 2010 Mar;16(3):265-73. doi: 10.1089/acm.2009.0399. PMID 20192911
- [Result] Brown R. Effects of Grounding on Body Voltage and Current in the Presence of Electromagnetic Fields. J Altern Complement Med. 2016 Sep;22(9):757-9. doi: 10.1089/acm.2015.0340. Epub 2016 Jul 25. PMID 27454187
- [Result] Brown R, Chevalier G, Hill M. Grounding after moderate eccentric contractions reduces muscle damage. Open Access J Sports Med. 2015 Sep 21;6:305-17. doi: 10.2147/OAJSM.S87970. eCollection 2015. PMID 26443876
- [Result] Chevalier G. Changes in pulse rate, respiratory rate, blood oxygenation, perfusion index, skin conductance, and their variability induced during and after grounding human subjects for 40 minutes. J Altern Complement Med. 2010 Jan;16(1):81-7. doi: 10.1089/acm.2009.0278. PMID 20064020
- [Result] Chevalier G. The effect of grounding the human body on mood. Psychol Rep. 2015 Apr;116(2):534-42. doi: 10.2466/06.PR0.116k21w5. Epub 2015 Mar 6. PMID 25748085
- [Result] Chevalier G, Patel S, Weiss L, Chopra D, Mills PJ. The Effects of Grounding (Earthing) on Bodyworkers' Pain and Overall Quality of Life: A Randomized Controlled Trial. Explore (NY). 2019 May-Jun;15(3):181-190. doi: 10.1016/j.explore.2018.10.001. Epub 2018 Oct 11. PMID 30448083
- [Result] Chevalier G, Sinatra ST, Oschman JL, Delany RM. Earthing (grounding) the human body reduces blood viscosity-a major factor in cardiovascular disease. J Altern Complement Med. 2013 Feb;19(2):102-10. doi: 10.1089/acm.2011.0820. Epub 2012 Jul 3. PMID 22757749
- [Result] Chevalier G, Sinatra ST, Oschman JL, Sokal K, Sokal P. Earthing: health implications of reconnecting the human body to the Earth's surface electrons. J Environ Public Health. 2012;2012:291541. doi: 10.1155/2012/291541. Epub 2012 Jan 12. PMID 22291721
- [Result] Cohen S, Janicki-Deverts D, Doyle WJ, Miller GE, Frank E, Rabin BS, Turner RB. Chronic stress, glucocorticoid receptor resistance, inflammation, and disease risk. Proc Natl Acad Sci U S A. 2012 Apr 17;109(16):5995-9. doi: 10.1073/pnas.1118355109. Epub 2012 Apr 2. PMID 22474371
- [Result] Elkin HK, Winter A. Grounding Patients With Hypertension Improves Blood Pressure: A Case History Series Study. Altern Ther Health Med. 2018 Nov;24(6):46-50. PMID 30982019
- [Result] Furman D, Campisi J, Verdin E, Carrera-Bastos P, Targ S, Franceschi C, Ferrucci L, Gilroy DW, Fasano A, Miller GW, Miller AH, Mantovani A, Weyand CM, Barzilai N, Goronzy JJ, Rando TA, Effros RB, Lucia A, Kleinstreuer N, Slavich GM. Chronic inflammation in the etiology of disease across the life span. Nat Med. 2019 Dec;25(12):1822-1832. doi: 10.1038/s41591-019-0675-0. Epub 2019 Dec 5. PMID 31806905
- [Result] Ghaly M, Teplitz D. The biologic effects of grounding the human body during sleep as measured by cortisol levels and subjective reporting of sleep, pain, and stress. J Altern Complement Med. 2004 Oct;10(5):767-76. doi: 10.1089/acm.2004.10.767. PMID 15650465
- [Result] Heneka MT, Carson MJ, El Khoury J, Landreth GE, Brosseron F, Feinstein DL, Jacobs AH, Wyss-Coray T, Vitorica J, Ransohoff RM, Herrup K, Frautschy SA, Finsen B, Brown GC, Verkhratsky A, Yamanaka K, Koistinaho J, Latz E, Halle A, Petzold GC, Town T, Morgan D, Shinohara ML, Perry VH, Holmes C, Bazan NG, Brooks DJ, Hunot S, Joseph B, Deigendesch N, Garaschuk O, Boddeke E, Dinarello CA, Breitner JC, Cole GM, Golenbock DT, Kummer MP. Neuroinflammation in Alzheimer's disease. Lancet Neurol. 2015 Apr;14(4):388-405. doi: 10.1016/S1474-4422(15)70016-5. PMID 25792098
- [Result] Johansson MM, Marcusson J, Wressle E. Cognitive impairment and its consequences in everyday life: experiences of people with mild cognitive impairment or mild dementia and their relatives. Int Psychogeriatr. 2015 Jun;27(6):949-58. doi: 10.1017/S1041610215000058. Epub 2015 Feb 3. PMID 25644289
- [Result] Kravitz BA, Corrada MM, Kawas CH. Elevated C-reactive protein levels are associated with prevalent dementia in the oldest-old. Alzheimers Dement. 2009 Jul;5(4):318-23. doi: 10.1016/j.jalz.2009.04.1230. PMID 19560102
- [Result] Lyra E Silva NM, Goncalves RA, Pascoal TA, Lima-Filho RAS, Resende EPF, Vieira ELM, Teixeira AL, de Souza LC, Peny JA, Fortuna JTS, Furigo IC, Hashiguchi D, Miya-Coreixas VS, Clarke JR, Abisambra JF, Longo BM, Donato J Jr, Fraser PE, Rosa-Neto P, Caramelli P, Ferreira ST, De Felice FG. Pro-inflammatory interleukin-6 signaling links cognitive impairments and peripheral metabolic alterations in Alzheimer's disease. Transl Psychiatry. 2021 Apr 28;11(1):251. doi: 10.1038/s41398-021-01349-z. PMID 33911072
- [Result] Menigoz W, Latz TT, Ely RA, Kamei C, Melvin G, Sinatra D. Integrative and lifestyle medicine strategies should include Earthing (grounding): Review of research evidence and clinical observations. Explore (NY). 2020 May-Jun;16(3):152-160. doi: 10.1016/j.explore.2019.10.005. Epub 2019 Nov 14. PMID 31831261
- [Result] Muller E, Proller P, Ferreira-Briza F, Aglas L, Stoggl T. Effectiveness of Grounded Sleeping on Recovery After Intensive Eccentric Muscle Loading. Front Physiol. 2019 Jan 28;10:35. doi: 10.3389/fphys.2019.00035. eCollection 2019. PMID 30745882
- [Result] Oschman JL, Chevalier G, Brown R. The effects of grounding (earthing) on inflammation, the immune response, wound healing, and prevention and treatment of chronic inflammatory and autoimmune diseases. J Inflamm Res. 2015 Mar 24;8:83-96. doi: 10.2147/JIR.S69656. eCollection 2015. PMID 25848315
- [Result] Oschman JL. Our place in nature: reconnecting with the Earth for better sleep. J Altern Complement Med. 2004 Oct;10(5):735-6. doi: 10.1089/acm.2004.10.735. No abstract available. PMID 15650460
- [Result] Oschman JL. Can electrons act as antioxidants? A review and commentary. J Altern Complement Med. 2007 Nov;13(9):955-67. doi: 10.1089/acm.2007.7048. PMID 18047442
- [Result] Oschman JL. Charge transfer in the living matrix. J Bodyw Mov Ther. 2009 Jul;13(3):215-28. doi: 10.1016/j.jbmt.2008.06.005. Epub 2008 Jul 30. PMID 19524846
- [Result] Oschman JL. Our place in nature: reconnecting with the Earth. J Altern Complement Med. 2010 Mar;16(3):225-6. doi: 10.1089/acm.2009.0656. No abstract available. PMID 20192906
- [Result] Oschman JL. Chronic disease: are we missing something? J Altern Complement Med. 2011 Apr;17(4):283-5. doi: 10.1089/acm.2011.0101. Epub 2011 Mar 25. No abstract available. PMID 21438673
- [Result] Passi R, Doheny KK, Gordin Y, Hinssen H, Palmer C. Electrical Grounding Improves Vagal Tone in Preterm Infants. Neonatology. 2017;112(2):187-192. doi: 10.1159/000475744. Epub 2017 Jun 10. PMID 28601861
- [Result] Pavlov VA, Tracey KJ. The vagus nerve and the inflammatory reflex--linking immunity and metabolism. Nat Rev Endocrinol. 2012 Dec;8(12):743-54. doi: 10.1038/nrendo.2012.189. PMID 23169440
- [Result] Sinatra ST, Oschman JL, Chevalier G, Sinatra D. Electric Nutrition: The Surprising Health and Healing Benefits of Biological Grounding (Earthing). Altern Ther Health Med. 2017 Sep;23(5):8-16. PMID 28987038
- [Result] Sokal K, Sokal P. Earthing the human body influences physiologic processes. J Altern Complement Med. 2011 Apr;17(4):301-8. doi: 10.1089/acm.2010.0687. Epub 2011 Apr 6. PMID 21469913
- [Result] Sokal K, Sokal P. Earthing the human organism influences bioelectrical processes. J Altern Complement Med. 2012 Mar;18(3):229-34. doi: 10.1089/acm.2010.0683. PMID 22420736
- [Result] Sokal P, Sokal K. The neuromodulative role of earthing. Med Hypotheses. 2011 Nov;77(5):824-6. doi: 10.1016/j.mehy.2011.07.046. PMID 21856083
- [Result] Thayer JF. Vagal tone and the inflammatory reflex. Cleve Clin J Med. 2009 Apr;76 Suppl 2:S23-6. doi: 10.3949/ccjm.76.s2.05. PMID 19376977
- [Result] Vinuesa A, Pomilio C, Gregosa A, Bentivegna M, Presa J, Bellotto M, Saravia F, Beauquis J. Inflammation and Insulin Resistance as Risk Factors and Potential Therapeutic Targets for Alzheimer's Disease. Front Neurosci. 2021 Apr 23;15:653651. doi: 10.3389/fnins.2021.653651. eCollection 2021. PMID 33967682
- [Result] Chevalier, G, & Sinatra, ST. Emotional Stress, Heart Rate Variability, Grounding, and Improved Autonomic Tone: Clinical Applications. Integrative Medicine. 2011; 10(3): 16-21.
- [Result] Chevalier, G, Melvin, G, & Barsotti, T. One-Hour Contact with the Earth's Surface (Grounding) Improves Inflammation and Blood Flow-A Randomized, Double-Blind, Pilot Study. Health. 2015; 07(08): 1022-1059.
- [Result] Chevalier, G. Grounding the human body improves facial blood flow regulation: Results of a randomized, placebo controlled pilot study. Journal of Cosmetics, Dermatological Sciences and Applications. 2014; 04(05): 293-308
- See also: "Beware of Misinformation" from The Earthing Institute — https://earthinginstitute.net/wp-content/uploads/2018/10/beware-of-earthing-misinformation-2018.pdf
- See also: "How to Measure the Effect of Earthing on Body Voltage" from The Earthing Institute — https://earthinginstitute.net/wp-content/uploads/2020/06/How-to-Measure-the-Effect-of-Earthing-on-Body-Voltage-2020.pdf
- See also: "Grounding Pain Patches: Every Medicine Cabinet Should Have Them" from The Earthing Institute — https://earthinginstitute.net/the-magic-pain-patches-every-medicine-cabinet-should-have-them/
- See also: "Medical and Medication Considerations" from The Earthing Institute — https://earthinginstitute.net/medical-and-medication-considerations/